CLINICAL TRIAL: NCT01731509
Title: "Early" Versus "Standard" Fetal Endoscopic Tracheal Occlusion for Severe Congenital Diaphragmatic Hernia - a Randomized Controlled Trial
Brief Title: Early FETO for Severe Congenital Diaphragmatic Hernia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8353/12
Record Dates: First submitted 2012-11-14; First posted 2012-11-21 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2012-11

CONDITIONS: Congenital Diaphragmatic Hernia
Keywords: congenital diaphragmatic hernia; fetoscopy; fetal endoscopic tracheal occlusion; pulmonary hypoplasia; fetal surgery; fetal lung
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard FETO (Active Comparator): Group of fetus that undergo fetal endoscopic tracheal occlusion between 26 0/7 weeks and 28 6/7 weeks.
  Interventions: Other: Fetal endoscopic tracheal occlusion
- Early FETO (Experimental): Group of fetus that undergo fetal endoscopic tracheal occlusion between 22 0/7 weeks and 24 6/7 weeks.
  Interventions: Other: Fetal endoscopic tracheal occlusion

INTERVENTIONS:
Other: Fetal endoscopic tracheal occlusion — FETO will be performed by placing a detachable balloon inside fetal trachea
  Other Names: FETO or fetal endoscopic traqueal occlusion

SUMMARY:
Congenital diaphragmatic hernia (CDH) is associated high mortality and morbidity, mainly in those cases with severe forms where there are extremely reduced lung volumes, liver herniation and decreased abnormal pulmonary vascularization. Fetal endoscopic tracheal occlusion performed between 26 and 30 weeks (standard FETO) has been shown to increase fetal pulmonary size and vascularity, and to improve infant survival in isolated severe CDH. Fetal pulmonary response followed FETO can be used to predict outcome and is dependent on the size of the fetal lung prior to the procedure.

We hypothesize that performing an earlier FETO, between 22-24 weeks, fetuses with severe form of CDH will have a better fetal pulmonary response and higher chance of surviving.

DETAILED DESCRIPTION:
We pretend to investigate if "early FETO" will improve the survival rate and the fetal pulmonary response, by conducting a randomized controlled trial comparing the results with those fetuses that undergo to "standard FETO" (between 26-28 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Fetuses with isolated congenital diaphragmatic hernia (normal fetal karyotype and absence of any associated structural anomaly);
* Gestational age established by last menstruation and/or first trimester ultrasonography;
* Prenatal diagnosis of congenital diaphragmatic hernia before 24 weeks of gestation
* Severe congenital diaphragmatic hernia (at 24 weeks, lung-to-head ratio <1.0 and at least 1/3 of the liver herniated into the fetal thorax)
* written informed consent (by the patient)

Exclusion Criteria:

* Preterm premature rupture of the membranes before randomization
* Preterm labor before randomization

Ages: 22 Weeks to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Infant survival rate | 6 months of life
  Percentage of survivors at 6 months of life

SECONDARY OUTCOMES:
Postnatal severe pulmonary arterial hypertension (PAH) | 30 days of life
  Severe PAH will be considered when the neonate presents with profound cyanosis associated with echocardiographic continuous right-to-left shunting through a persistent 'ductus arteriosus' and a persistent difference in pre- to postductal saturation gradient >20%, despite the use of intake Nitric Oxide (iNO).
Respiratory morbidity | 6 months of life
  Need for ventilatory support and/or oxygen dependency.

OTHER OUTCOMES:
obstetrical complications (morbidity) | pregnancy
  1. Preterm premature rupture of the membranes (<37 weeks)
  2. Extremely preterm premature rupture of the membranes (<32 weeks)
  3. Preterm delivery (birth <37 weeks of gestation)
  4. Extremely preterm delivery (birth <32 weeks)
  5. Placental abruption
  6. Chorioamnionitis and maternal infection

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Ruano, MD PhD, Principal Investigator — Faculdade de Medicina da Universidade de Sao Paulo
Locations (1):
- Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Ruano R, Duarte SA, Pimenta EJ, Takashi E, da Silva MM, Tannuri U, Zugaib M. Comparison between fetal endoscopic tracheal occlusion using a 1.0-mm fetoscope and prenatal expectant management in severe congenital diaphragmatic hernia. Fetal Diagn Ther. 2011;29(1):64-70. doi: 10.1159/000311944. Epub 2010 Apr 10. PMID 20389048
- [Background] Ruano R, Yoshisaki CT, da Silva MM, Ceccon ME, Grasi MS, Tannuri U, Zugaib M. A randomized controlled trial of fetal endoscopic tracheal occlusion versus postnatal management of severe isolated congenital diaphragmatic hernia. Ultrasound Obstet Gynecol. 2012 Jan;39(1):20-7. doi: 10.1002/uog.10142. Epub 2011 Dec 14. PMID 22170862
- [Background] Ruano R, da Silva MM, Campos JA, Papanna R, Moise K Jr, Tannuri U, Zugaib M. Fetal pulmonary response after fetoscopic tracheal occlusion for severe isolated congenital diaphragmatic hernia. Obstet Gynecol. 2012 Jan;119(1):93-101. doi: 10.1097/AOG.0b013e31823d3aea. PMID 22183216
- [Background] Harrison MR, Keller RL, Hawgood SB, Kitterman JA, Sandberg PL, Farmer DL, Lee H, Filly RA, Farrell JA, Albanese CT. A randomized trial of fetal endoscopic tracheal occlusion for severe fetal congenital diaphragmatic hernia. N Engl J Med. 2003 Nov 13;349(20):1916-24. doi: 10.1056/NEJMoa035005. PMID 14614166
- [Background] Jani JC, Nicolaides KH, Gratacos E, Valencia CM, Done E, Martinez JM, Gucciardo L, Cruz R, Deprest JA. Severe diaphragmatic hernia treated by fetal endoscopic tracheal occlusion. Ultrasound Obstet Gynecol. 2009 Sep;34(3):304-10. doi: 10.1002/uog.6450. PMID 19658113
- [Background] Deprest J, Gratacos E, Nicolaides KH; FETO Task Group. Fetoscopic tracheal occlusion (FETO) for severe congenital diaphragmatic hernia: evolution of a technique and preliminary results. Ultrasound Obstet Gynecol. 2004 Aug;24(2):121-6. doi: 10.1002/uog.1711. PMID 15287047